CLINICAL TRIAL: NCT06309472
Title: A Multi-centre, Double-blind Randomised Controlled Trial to Compare Mirtazapine Versus Placebo Over 12 Weeks in Patients With Multimorbid Major Depression and Inflammatory Bowel Disease (MD-IBD): a Feasibility Study
Brief Title: Trial of Mirtazapine for Depression in IBD
Acronym: MDIBD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: King's College Hospital NHS Trust (Other); Imperial College London (Other); London North West Healthcare NHS Trust (Other); Imperial College Healthcare NHS Trust (Other); Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Calum Moulton, Chief Investigator, King's College London
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIHR302528
Record Dates: First submitted 2024-02-27; First posted 2024-03-13 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Major Depressive Disorder; Inflammatory Bowel Diseases
Keywords: Mirtazapine; Placebo; Depression; Randomised controlled trial; Feasibility trial; Inflammatory bowel disease; Crohn's disease; Ulcerative colitis
MeSH Terms: conditions — Depressive Disorder, Major; Inflammatory Bowel Diseases; Depression; Crohn Disease; Colitis, Ulcerative | interventions — Mirtazapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Mirtazapine and placebo manufactured to appear identical through over-encapsulation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirtazapine (Experimental): Mirtazapine 30-45mg at night for 12 weeks
  Interventions: Drug: Mirtazapine
- Placebo (Placebo Comparator): Matched placebo 1-2 capsules at night for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mirtazapine — 30mg mirtazapine at night, escalated to 45mg after 4 weeks if <20 percent improvement in depression from baseline. Total treatment duration 12 weeks.
  Other Names: Remeron
  Arms: Mirtazapine
Drug: Placebo — 1 placebo capsule at night, escalated to 2 capsules after 4 weeks if <20 percent improvement in depression from baseline. Total treatment duration 12 weeks.
  Arms: Placebo

SUMMARY:
This study will test whether it is feasible to conduct a clinical trial of mirtazapine (an antidepressant tablet) in patients who have both depression and inflammatory bowel disease (IBD). The study design is a randomised controlled trial (a study in which people are allocated by chance to receive different interventions). The trial will compare mirtazapine against a placebo (dummy) tablet in 76 patients with both depression and IBD.

The investigators will recruit outpatients aged 18 or over with a diagnosis of any IBD attending gastroenterology clinics. Either in person or remotely, patients will complete a brief screening questionnaire for depression. Those scoring positive for depression will be invited for a 15-minute interview for clinical depression. Those with clinical depression will be invited to take part. Participants will be randomly allocated by a computer to take either 1) mirtazapine tablet once at night for 12 weeks; or 2) placebo (dummy) tablet once at night for 12 weeks. The study is 'blinded', meaning neither patients nor the study team will know which medication they are taking. Throughout, participants will be able to access other treatments for depression, such as talking therapies.

The investigators will measure how many people join the study; how many remain in the trial; how many complete treatment; how many tablets people take; and assess overall acceptability of the trial. Participants will complete brief questionnaires to measure their mental health and IBD symptoms after 4 weeks, 8 weeks, 12 weeks and 16 weeks. Participants will also provide blood samples and faecal samples to measure inflammation.

If successful, this trial will support an application for a larger version of the study.

DETAILED DESCRIPTION:
Background:

Depression is highly prevalent in patients with inflammatory bowel disease (IBD) and associated with poor IBD outcomes. Mirtazapine, a tetracyclic antidepressant, is particularly promising in IBD because it has minimal effect on gut motility; has anti-emetic effects; is well absorbed from the gut and carries a low risk of sexual dysfunction. However, mirtazapine has never been trialed in patients with IBD.

Aim:

To test whether it is feasible to carry out a trial of mirtazapine versus placebo - both in addition to treatment-as-usual - for the treatment of depression in patients with IBD, in order to inform the design of a subsequent powered multi-centre randomised controlled trial (RCT).

Objectives:

The primary aim of the research is to test the feasibility of a definitive trial of mirtazapine + treatment-as-usual (TAU) against matched placebo + TAU for depression in adults with IBD. This study will:

1. Establish recruitment, retention, and adherence rates
2. Measure acceptability using treatment adherence and qualitative interview
3. Test the assessment methods and procedures for measuring variables for use in a full trial
4. Test the feasibility of collecting health economic data, including health service use

   Study design:

   The study is a parallel group, 1:1 feasibility randomised controlled trial (RCT). Participants will be randomised to one of the two treatment arms (mirtazapine + treatment-as-usual (TAU) or matched placebo + TAU) and will complete measures at baseline, 4 weeks, 8 weeks and 12-weeks post randomisation. Blinded treatment will last for 12 weeks, followed by the offer of a 2-3-week tapering off dose. A post-treatment follow-up will take place at 16 weeks post-randomisation.

   Recruitment:

   From outpatient gastroenterology services, patients aged ≥18 and diagnosed with Crohn's disease or ulcerative colitis, confirmed using clinical notes, will be screened for depression using the Patient Health Questionnaire-9 (PHQ-9) as part of clinical care. For those with at least moderate depression (≥10 on the PHQ-9) - the clinical team will seek the patient's permission to be contacted by the research team. Those who are deemed to be potentially eligible will be invited for a screening assessment with a member of the study team. Final study inclusion and consent will be taken by a member of the study team.

   Assignment of interventions:

   Participants will be randomly assigned to either mirtazapine or placebo with a 1:1 allocation as per a computer-generated randomisation schedule, which will use a varying permuted block design stratified by diagnosis (Crohn's disease or ulcerative colitis) and sex assigned at birth (male/female). The block sizes will not be disclosed. Participants will be randomised by the clinical team using a web based online randomisation system.

   Blinding:

   Participants and researchers will be blind to treatment allocation. The blinding will be maintained by opaque over-encapsulation of mirtazapine/placebo. Assessments regarding clinical outcomes will be conducted by an assessor blind to treatment allocation. The trial statistician will become unblind after the first version of the Statistical Analysis Plan is signed.

   Intervention:

   Half (n=38) will be randomised to 12 weeks of treatment with mirtazapine, which will be blinded through over-encapsulation. The starting dose will be 30mg once at night (ON), which is the minimum therapeutic dose for depression. Treatment with mirtazapine will occur in addition to treatment-as-usual, which is any psychological therapy the patient wishes to access through the National Health Service (NHS) or private therapy services. The patient and assessor will remain blinded to treatment allocation throughout the 12 weeks of treatment. Most benefit from antidepressants is gained within the first 2 weeks after starting treatment, and 12 weeks is a standard treatment duration for antidepressant trials.

   After 4 weeks of taking mirtazapine 30mg at night, clinical response will be assessed using the Quick Inventory for Depressive Symptomatology-16. In accordance with British Association of Psychopharmacology clinical guidelines, the dose will be increased to 45mg at night if there is <20 percent clinical improvement from baseline.

   The other half (n=38) will be randomised to a matched placebo, which is a matched capsule filled with lactose. Treatment with placebo will occur in addition to treatment-as-usual, which is any psychological therapy the patient wishes to access through NHS services or private therapy services. After 4 weeks of taking placebo 1 capsule at night, clinical response will be assessed using the Quick Inventory for Depressive Symptomatology-16. The dose will be increased to 2 capsules at night if there is <20 percent clinical improvement from baseline.

   Continuity of care:

   The investigators will ask participants if they wish to continue mirtazapine through their General Practitioner (GP) after their participation in the trial has finished. For those not wishing to continue treatment after the trial, participants will be able to down-titrate and stop treatment.

   Concomitant medications:

   Participants will agree not to start any other antidepressants during the trial. The investigators will also exclude participants where there is a planned or expected change in IBD treatment in the next 12 weeks. The investigators will record concomitant medications for IBD, mental health or pain (strong or weak opioids) during this time.

   Treatment stopping rules:

   Treatment will be stopped for an individual participant if they develop any of the following:
   * Active suicidal thoughts.
   * Pregnancy
   * Any Serious Adverse Event (SAE), Serious Adverse Reaction (SAR) or Unexpected Serious Adverse Reaction (USAR), which, in the view of the investigators, necessitates treatment cessation.

   Every effort will be made to ensure the patient outcomes are continued to be collected even if their treatment has been stopped.

   Withdrawal:

   Participants have the right to withdraw from the study at any time for any reason. The investigators also have the right to withdraw participants from the study in the event of inter-current illness, adverse events, protocol or treatment non-compliance or administrative reasons. Should a participant withdraw from the intervention, efforts will be made to continue to obtain follow-up data, with the permission of the patient.

   Measures collected at baseline:

   Socio-demographic variables: age, sex, ethnicity, occupational status, duration of education, marital status, current employment status and smoking status.

   Psychiatric history: previous episodes of depression or anxiety, medication history, previous psychological therapies and psychiatric comorbidities.

   IBD variables: IBD diagnosis, disease type using the Montreal classification, IBD duration, current/previous medications, current analgesia, presence/absence of fistulae, current stoma (colostomy, ileostomy, jejunostomy), current or previous parenteral nutrition or intravenous fluid support, previous surgery and number of IBD flares in the last 2 years.

   Anthropometrics: Height and weight for participants attending in person.

   Primary feasibility outcomes:

   These are described in detail elsewhere.

   Secondary outcomes (baseline, 4 weeks, 8 weeks, 12 weeks and 16 weeks post-randomisation):

   Participants will complete a questionnaire schedule that includes key psychological measures, typically completed within 30 minutes by patients themselves. The investigators will repeat the range of questionnaires at follow-up and estimate the completeness, variance and estimate standardised effect sizes (see Outcomes section), as well as faecal calprotectin, C-reactive protein and inflammatory cytokines. Effects on gut microbiome, gut metabolome and serum metabolome will also be captured and reported outside of the main trial analysis.

   Qualitative interview (subset of participants, after completion of the trial):

   We will also assess feasibility using a one-off post-treatment interview, conducted between 12- and 16 weeks after initial randomisation. The investigators will approach all patients who begin treatment but discontinue, exploring their reasons and any barriers they encountered. A purposive sample of treatment completers will also be invited to individual post-treatment interviews.

   End of study definition:

   The end of the trial will be defined as the date when all participants have made their final visits, the data entered into the database and all queries resolved and the database locked.

   Sample size:

   As a feasibility study, power calculations for a treatment effect are not applicable. The target sample size is 64 participants (32 per group), which is sufficient to generate robust variance estimates. To account for an estimated 15% attrition, the investigators will recruit 76 participants to the study. Based on this sample size, a two-sided confidence interval will extend no more than 10% of the observed proportion.

   Data management:

   Data will be collected on paper case report form (CRF) and then transferred to an electronic case report form (eCRF). The type of activity that an individual user may undertake is regulated by the privileges associated with his/her user identification code and password. All forms and tapes related to study data will be kept in locked cabinets. Access to the study data will be restricted. The database will be password-protected.

   Statistical methods:

   A statistical analysis plan (SAP) will be approved by the Trial Steering Committee independent statistician. The analysis population will use intention-to-treat principles. A recruitment plot of predicted vs. actual recruitment will be generated on a monthly basis.

   Participant flow through the study will be presented. Descriptive data will be presented in the form of means and standard deviations; medians and ranges; or percentages with 95% confidence intervals, as appropriate depending on the data being described. The investigators will use linear mixed models to estimate the between group adjusted mean difference (aMD) between mirtazapine and placebo groups at week 12 after adjustment for baseline scores, time, and a treatment-by-time-interaction. Associated 95% confidence intervals will be presented alongside the aMD without p-values. More details will be provided in the statistical analysis plan.

   Exploratory analysis:

   To explore potential mediators of treatment response in a future powered trial (reduction in peripheral inflammatory cytokines, improvement in sleep quality, improvement in irritable bowel syndrome symptoms, improvement in functional dyspepsia symptoms), exploratory analysis will report the mediation analysis. Significant findings will be interpreted cautiously, acknowledging the issue of multiple testing, need for replication and low statistical power.

   Qualitative data analysis:

   For the qualitative analysis of post-treatment interviews, the investigators will use pragmatic thematic analysis to code and report the interview data. Two researchers will perform preliminary analysis to identify themes, which will then be discussed and agreed with all authors if appropriate.

   Dissemination policy:

   Findings of this feasibility study will be disseminated through international conferences, peer-reviewed journals, charities, educational seminars in acute trusts and through appropriate social media channels. If the study is feasible, it will support an application for a powered trial of mirtazapine for depression in IBD.

ELIGIBILITY:
Inclusion Criteria:

1. Established diagnosis of Crohn's disease (CD) or ulcerative colitis (UC) according to clinical notes
2. Fulfil Diagnostic and Statistical Manual of Mental Disorders (5th Edition) (DSM-5) criteria for current single or recurrent episodes of major depressive disorder of at least moderate severity but without psychotic features, as defined by the Mini Neuropsychiatric Interview
3. Aged 18 years or over
4. Use of contraception if female and of childbearing age. Female participants of childbearing age will require a negative serum/urine pregnancy test before starting the study and will also need to agree to use an acceptable form of contraception throughout the intervention period, e.g. oral contraceptive pill, long-acting reversible contraceptive
5. Able to provide written informed consent to enter the trial

Exclusion Criteria:

1. Diagnosis of drug or alcohol dependence syndrome according to the General Practitioner (GP) summary care record or yes in answer to the question "have you ever been diagnosed with drug or alcohol dependence?"
2. Diagnosis of any personality disorder according to the GP summary care record or yes in answer to the question "have you ever been diagnosed with a personality disorder?"
3. Diagnosis of any dementia according to the GP summary care record or yes in answer to the question "have you ever been diagnosed with any form of dementia?"
4. Diagnosis of psychosis or schizophrenia according to the GP summary care record or yes in answer to the question "have you ever been diagnosed with psychosis or schizophrenia?"
5. Diagnosis of bipolar disorder according to the GP summary care record or yes in answer to the question "have you ever been diagnosed with bipolar disorder?"
6. Current active suicidal ideation on clinical assessment according to clinical judgment by a study consultant psychiatrist
7. Current treatment with mirtazapine, mianserin, trazodone or a monoamine oxidase inhibitor
8. Contraindications to the administration of mirtazapine, as per the current summary of product characteristics
9. Known allergy to mirtazapine or mianserin according to patient report or clinical notes
10. Non-registration with a GP or failure to consent to sharing of the GP summary care record and any psychiatric assessments held
11. Currently enrolled in another drug trial or psychological therapy trial
12. Currently hospitalised for the treatment of IBD
13. Currently being prescribed a course of budesonide or reducing course of prednisolone for IBD
14. Planned change in IBD treatment within the next 12 weeks according to clinical notes or answer yes to the question: "are you expecting any change in your IBD treatment to take place in the next 12 weeks?"

Ages: 18 Years to 125 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Recruitment feasibility | Up to 2 years
  Participants randomised overall, percentage of target
Trial adherence | 12 weeks
  Percentage of participants completing 12 weeks of treatment
Treatment adherence | 12 weeks
  Percentage of participants taking at least 75% of prescribed mediation
Study procedures acceptability and compliance | 12 weeks
  Percentage of planned data and samples collected at primary endpoint (12 weeks)
Overall acceptability | 12 weeks
  Percentage of participants describing the treatment as acceptable (≥6/10 on 0-10 scale)

SECONDARY OUTCOMES:
Quick Inventory for Depressive Symptomatology-16 Questionnaire | Baseline, 4, 8, 12 and 16 weeks
  Range 0-27, higher scores indicate worse depressive symptoms
Patient Health Questionnaire-9 questionnaire | Baseline, 4, 8, 12 and 16 weeks
  Range 0-27, higher scores indicate worse depressive symptoms
Generalised Anxiety Disorder-7 questionnaire | Baseline, 4, 8, 12 and 16 weeks
  Range 0-21, higher scores indicate worse anxiety symptoms
Inflammatory Bowel Disease Control questionnaire | Baseline, 4, 8, 12 and 16 weeks
  Range 0-16, higher scores indicate better self-report IBD control
Inflammatory Bowel Disease Fatigue Assessment Scale | Baseline, 4, 8, 12 and 16 weeks
  Range 0-20, higher scores indicate worse fatigue severity
Chalder Fatigue Scale | Baseline, 4, 8, 12 and 16 weeks
  Range 0-11, higher scores indicate worse fatigue severity
Maudsley 3-item Visual Analogue Scale | Baseline, 4, 8, 12 and 16 weeks
  Range 0-300, higher scores indicate worse depressive symptoms
Pittsburgh Sleep Quality Index | 4, 8, 12 and 16 weeks
  Range 0-21, higher scores indicate worse sleep
9-item Avoidant Restrictive Food Intake Disorder Screen | Baseline, 4, 8, 12 and 16 weeks
  Range 0-45, higher scores indicate worse symptoms
Patient Assessment of Gastrointestinal Disorders Symptom Severity Index (PAGI-SYM) Questionnaire | Baseline, 4, 8, 12 and 16 weeks
  Range 0-100, higher scores indicate worse gastrointestinal symptoms
Inflammatory Bowel Disease Resource Use Questionnaire (IBD-RUQ) items on employment and healthcare contacts | Baseline, 4, 8, 12 and 16 weeks
  Higher number of healthcare contacts indicates worse outcome. No minimum or maximum values
Birmingham Irritable Bowel Syndrome Symptoms Questionnaire | Baseline, 4, 8, 12 and 16 weeks
  Range 0-55, higher scores indicate worse symptoms
Harvey Bradshaw Index (Crohn's disease patients only) | Baseline and 12 weeks
  No upper limit. Higher scores indicate worse disease, specifically: Remission: <5, Mild Disease: 5-7, Moderate Disease: 8-16, Severe Disease: >16
Simple Clinical Colitis Activity Index (ulcerative colitis patients only) | Baseline and 12 weeks
  Range 0-19, higher scores indicate worse symptoms
Dietary Screener Questionnaire | Baseline and 12 weeks
  No maximum value, higher scores indicate increased dietary content
Concentration of faecal calprotectin | Baseline and 12 weeks
  Range 5-8000, higher scores suggest worse disease activity
Concentration of serum high-sensitivity C-reactive protein | Baseline and 12 weeks
  Range 1-400, higher scores indicate elevated inflammatory activity
Concentration of serum interleukin-23 | Baseline and 12 weeks
  Range 6.8-2500, higher scores indicate elevated inflammatory activity
Concentration of serum interleukin-22 | Baseline and 12 weeks
  Range 16.6-63300, higher scores indicate elevated inflammatory activity
Concentration of serum granulocyte-macrophage colony-stimulating factor | Baseline and 12 weeks
  Range 1.4-13460, higher scores indicate elevated inflammatory activity
Concentration of serum interleukin-5 | Baseline and 12 weeks
  Range 0.26-2496, higher scores indicate elevated inflammatory activity
Concentration of serum interleukin-13 | Baseline and 12 weeks
  Range 7.2-27440, higher scores indicate elevated inflammatory activity
Concentration of serum interleukin-17A | Baseline and 12 weeks
  Range 2.1-20000, higher scores indicate elevated inflammatory activity
Concentration of serum tumor necrosis factor alpha | Baseline and 12 weeks
  Range 0.6-2320, higher scores indicate elevated inflammatory activity
Concentration of serum interferon-gamma | Baseline and 12 weeks
  Range 0.34-8000, higher scores indicate elevated inflammatory activity

CONTACTS AND LOCATIONS:
Overall Officials: Calum D Moulton, PhD, Principal Investigator — King's College London
Locations (4):
- United Kingdom (4):
  - Guy's and St Thomas' Hospital NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - King's College Hospital NHS Foundation Trust, London
  - St Mark's Hospital, London

IPD SHARING:
Plan to Share IPD: No